CLINICAL TRIAL: NCT02067832
Title: Applying Biomarkers to Long-term Effects in Child and Adolescent Cancer Treatment (ABLE Team) - Predictive Biomarkers For Pediatric Chronic Graft-Versus-Host Disease
Brief Title: Predictive Biomarkers For Pediatric Chronic Graft-Versus-Host Disease
Acronym: ABLE-cGVHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kirk Schultz, Principle Investigator, University of British Columbia
Other Study IDs: H12-02890; TCF-118695 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2014-01-20; First posted 2014-02-20 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Chronic Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — From recipient: whole blood From donor: bone marrow or apheresis product
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic graft-versus-host disease (cGVHD) can be hard to diagnose, difficult to manage and contributes significantly to morbidity and mortality in hematopoietic stem cell transplantation patients.

The research will look into identifying and validating cGVHD biological indicators (=bio-markers) which will be evaluated whether they can predict a future development of the disease.

The study hypothesis is that a number of previously reported cGVHD bio-markers, known to be present at the time of cGVHD diagnosis, will also be present at earlier time points, before cGVHD develops.

Following validation, the bio-markers will be beneficial for finding those patients who are in higher risk to develop cGVHD.

By identifying the higher-risk group, which is more likely to develop cGVHD, a pre-emptive therapy might be applied in order to prevent or reduce the prevalence of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Allogeneic hematopoietic stem cell transplantation for any malignant or non-malignant disease.
2. Age 0-17.99 years at the time of transplantation.
3. Bone marrow, peripheral blood stem cell and umbilical cord blood (including single or double cord blood) as the graft source.
4. Any conditioning regimen with any chemotherapy / radiation therapy combination. Haploidentical donor transplants with post-transplant cyclophosphamide are also allowed.
5. Use of serotherapy is permitted.
6. Any graft-versus-host disease prophylaxis is permitted, including post-HSCT cyclophosphamide.
7. If participant weighs between 0-20 kg, participant must be able to provide 15 ml of whole blood at each time point.
8. If participant weighs over 20 kg, participant must be able to provide 1ml/kg of whole blood, up to a maximum of 23 mL for the pre-conditioning sample and 32 mL for samples at day +100, 6-months, 12-months, +/- the cGVHD sample.
9. Written informed consent from parents.
10. Assent from study participant when appropriate.
11. Participation on other clinical trials is acceptable.

Exclusion Criteria:

1. Autologous HSCT.
2. Patients referred to a Bone Marrow Transplant (BMT) center from a non-BMT center, where it is anticipated (at the discretion of the center PI) that adequate follow up according to the rules of this protocol can not be met, including the requirement for a reassessment by the BMT center at the time of cGVHD diagnosis.
3. Ex-vivo T-cell depletion of graft source (e.g. CD34 selection).
4. Second (or greater) allogeneic transplants (first allogeneic transplant where a previous autologous transplant was performed is permitted).
5. Syngeneic transplants.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Recipients and donors of allogeneic hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive bio-markers for pediatric chronic Graft-Versus-Host Disease (cGVHD) in Hematopoietic Stem Cell Transplant (HSCT) recipients | Just before transplant to 12 months post transplant or until diagnosis of cGVHD if precede the 12 months
  The study will try to determine the prevalence (or levels) of high-probability predictive plasma and cellular cGVHD bio-markers in pediatric patients undergoing allogeneic HSCT from blood samples

SECONDARY OUTCOMES:
Validation of "predictive" cGVHD bio-markers | Measure will be assessed following the submission of all samples. During the last year of the study (Oct. 2016 - Sept. 2017)
  To determine and validate whether "predictive" cGVHD bio-markers present before the onset of cGVHD are able to predict a subset of pediatric patients at greatest risk for the development of cGVHD in the future

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Cuvelier, MD, Principal Investigator — University of Manitoba; Kirk R Schultz, MD, Principal Investigator — University of British Columbia
Locations (25):
- United States (18):
  - Children's of Alabama, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Nemours A. I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - C S Mott Children's Hospital The University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Blair E. Batson Hospital for Children, Jackson, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morgan Stanley Children's Hospital, New York, New York
  - New York Medical College, Valhalla, New York
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Utah Primary Children's Medical Center, Salt Lake City, Utah
- ST.Anna Children's Hospital, Vienna, Austria
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of British Columbia - BC Children's Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - The Sainte-Justine University Hospital Centre, Montreal, Quebec

REFERENCES:
- [Derived] Cuvelier GDE, Ng B, Abdossamadi S, Nemecek ER, Melton A, Kitko CL, Lewis VA, Schechter T, Jacobsohn DA, Harris AC, Pulsipher MA, Bittencourt H, Choi SW, Caywood EH, Kasow KA, Bhatia M, Oshrine BR, Chaudhury S, Coulter D, Chewning JH, Joyce M, Savasan S, Pawlowska AB, Megason GC, Mitchell D, Cheerva AC, Lawitschka A, Ostroumov E, Schultz KR. A diagnostic classifier for pediatric chronic graft-versus-host disease: results of the ABLE/PBMTC 1202 study. Blood Adv. 2023 Jul 25;7(14):3612-3623. doi: 10.1182/bloodadvances.2022007715. PMID 36219586
- [Derived] Subburaj D, Ng B, Kariminia A, Abdossamadi S, Lauener M, Nemecek ER, Rozmus J, Kharbanda S, Kitko CL, Lewis VA, Schechter-Finklestein T, Jacobsohn DA, Harris AC, Pulsipher MA, Bittencourt H, Choi SW, Caywood EH, Kasow KA, Bhatia M, Oshrine BR, Coulter D, Chewning JH, Joyce M, Pawlowska AB, Megason GC, Lawitschka A, Ostroumov E, Klein Geltink R, Cuvelier GDE, Schultz KR. Metabolomic identification of alpha-ketoglutaric acid elevation in pediatric chronic graft-versus-host disease. Blood. 2022 Jan 13;139(2):287-299. doi: 10.1182/blood.2021013244. PMID 34534280